CLINICAL TRIAL: NCT06682143
Title: The Effects of Virtual Reality Greenspace Exposure on Physiological and Affective Acute Stress Responses Among Adults With Mobility Impairments: A Pilot Study
Brief Title: The Effects of Virtual Reality Greenspace on Stress Among Adults With Mobility Impairments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Laurie A Malone, PhD, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300012947
Record Dates: First submitted 2024-10-22; First posted 2024-11-12 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Mobility Impairments
Keywords: stress; mobility impairment; virtual reality; greenspace

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): Participants will be outfitted with a virtual reality headset. While seated in a recliner chair, participants will engage in a pre-specified VR nature experience called Nature Treks VR for 5 minutes.
  Interventions: Behavioral: Virtual Reality (VR)
- Control (Placebo Comparator): Participants will be seated in a recliner chair and asked to sit quietly for 5 minutes.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Virtual Reality (VR) — Participants will engage in a virtual reality greenspace activity for a period of 5 minutes
  Arms: Virtual reality
Behavioral: Control — Participants will sit quietly for a period of 5 minutes
  Arms: Control

SUMMARY:
The purpose of this project is to examine the effects of virtual reality greenspace exposure on physiological and affective acute stress responses among adults with mobility impairments.

DETAILED DESCRIPTION:
Exposure to greenspace is known to yield numerous mental and physical health benefits such as improved mood, decreased stress, and increased levels of physical activity. Regular access to greenspace however is difficult for various segments of the population including individuals with disabilities or chronic health conditions. Numerous factors contribute to this difficulty including architectural barriers, shortage of accessible trails, and limited transportation options. These challenges have led to a growing interest in exploring the use of virtual reality (VR) greenspace environments. Studies have demonstrated that VR greenspace exposure can reduce stress and improve mood and mental well-being in various populations but has not been tested among individuals with mobility impairments who experience high levels of stress. During a single lab visit, participants will be randomized to VR greenspace activity or control, undergo the Trier Social Stress Test. The VR group will then engage in a series of nature-based VR activities. The Control group will sit quietly. Assessments will be collected at 4 timepoints. Physiological stress responses will be measured via changes in BP, HR, and two saliva measures (salivary alpha-amylase, salivary cortisol). Affective response (stress, affect, anxiety) will be assessed using self-report surveys. This study will provide insight into the influence of VR greenspace exposure on stress recovery (physiological and affective responses), among individuals with mobility impairments.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* A self-reported lower extremity mobility impairment (e.g., cerebral palsy, spinal cord injury, multiple sclerosis, stroke) with partial or full use of the upper extremities.

Exclusion Criteria:

* Impairment in visual acuity as measured by a Snellen eye chart <20/70 after correction
* Regular engagement (>20 minutes/week) in virtual reality greenspace activity
* Having an endocrine disorder (that can affect cortisol levels)
* Taking oral corticosteroids
* Score below 24 on the Mini Mental State Exam

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | The survey will be completed at 4 timepoints: 1) Baseline (Stage 1) 2) Immediately after the Trier Social Stress Test (Stage 2); 3) Immediately following the VR or control activity; 4) 20 minutes after completion of the activity (VR or control).
  The survey consists of 10 questions that assess the frequency of feelings and thoughts related to stress on a 5-point Likert scale (Never = 0, Almost never = 1, Sometimes = 2, Fairly often = 3; Very often = 4). To calculate a total PSS score, responses to the four positively stated items (items 4, 5, 7 and 8) first need to be reversed (i.e. 0 => 4; 1 => 3; 2 => 2; 3 => 1; 4 => 0). The PSS score is then obtained by summing across all items. Higher scores indicate higher levels of perceived stress.
State-Trait Anxiety Inventory (STAI) short form | The survey will be completed at 4 timepoints: 1) Baseline (Stage 1); 2) Immediately after the Trier Social Stress Test (Stage 2); 3) Immediately following the VR or control activity; 4) 20 minutes after completion of the activity (VR or control).
  The 5-item short form of the State-Trait Anxiety Inventory (STAI) is designed to quickly assess anxiety levels. The questions measure state (temporary feelings of anxiety) and trait anxiety (general tendency to experience anxiety).The STAI short form is scored by summing the responses to each of the five items, which are rated on a 4-point Likert scale ranging from 1 (not at all) to 4 (very much so). The total score can range from 5 to 20, with higher scores indicating higher levels of anxiety.
Positive and Negative Affect Schedule | The survey will be completed at 4 timepoints: 1) Baseline (Stage 1); 2) Immediately after the Trier Social Stress Test (Stage 2); 3) Immediately following the VR or control activity; 4) 20 minutes after completion of the activity (VR or control).
  The Positive and Negative Affect Schedule (PANAS) is designed to measure positive and negative affect. It consists of 20 items, with 10 items each for positive affect (PA) and negative affect (NA). Respondents rate each item on a 5-point Likert scale ranging from 1 (very slightly or not at all) to 5 (extremely). Positive Affect Score: Sum the scores of items 1, 3, 5, 9, 10, 12, 14, 16, 17, and 19. Scores can range from 10 to 50, with higher scores indicating higher levels of positive affect. Negative Affect Score: Sum the scores of items 2, 4, 6, 7, 8, 11, 13, 15, 18, and 20. Scores can range from 10 to 50, with higher scores indicating higher levels of negative affect.
Saliva stress biomarkers | The saliva will be collected at 4 timepoints: 1) Baseline (Stage 1); 2) Immediately after the Trier Social Stress Test (Stage 2); 3) Immediately following the VR or control activity; 4) 20 minutes after completion of the activity (VR or control).
  Saliva samples will be collected to measure stress biomarkers. The process is simple and non-invasive:
  Preparation: Participants should avoid eating, drinking (except water), brushing teeth, or using mouthwash for at least 30 minutes before sample collection.
  Collection: Participants will be provided with a sterile saliva collection device. They will be asked to spit into the device until it reaches the indicated fill line.
  Storage: The collected saliva samples will be stored in a cooler bag and then later transported to the UAB lab for storage and analyses.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study so IPD will not be shared.